CLINICAL TRIAL: NCT01598740
Title: A Phase 1, Open-label, Randomized, Crossover Study to Assess the Safety, Tolerability, and Efficacy of CLP With and Without Spironolactone in Adults With Heart Failure
Brief Title: Evaluation of CLP With and Without Spironolactone in Heart Failure Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorbent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTST-25
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLP with spironolactone (Experimental)
  Interventions: Drug: CLP; Drug: Spironolactone
- CLP without spironolactone (Experimental)
  Interventions: Drug: CLP

INTERVENTIONS:
Drug: CLP — Oral administration
Drug: Spironolactone — oral administration
  Arms: CLP with spironolactone

SUMMARY:
The purpose of this study is to determine the effects of CLP, with and without spironolactone, on serum, urine, and fecal contents in heart failure patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with New York Heart Association (NYHA) Classification II or III
* Chronic kidney disease
* Cardiac ejection fraction <40%
* On heart failure therapy including an ACEI or ARB, and a BB
* Willing to understand and comply with study procedures and provide written informed consent.

Exclusion Criteria:

* Hospitalization within 4 weeks of baseline visit
* History or presence of gastrointestinal conditions such as severe constipation or gastrointestinal tract strictures
* Current or anticipated dialysis during study
* In the investigator's judgment, any cardiovascular, renal, hepatic, endocrine, gastrointestinal, neurological, or other disease or condition that makes the subject's study participation unsafe
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dittrich, MD, Study Chair — Sorbent Therapeutics, Study Sponsor; Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange Country Research Center, Tustin, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 01 June 2012 and the last subject completed on 06 August 2012. The study was completed at one research center.
Pre-assignment Details: Each study period included a 5-day baseline period followed by a 7-day treatment period. The study periods were separated by a 7-day washout period.
Groups:
- CLP + Spiro (7 Days), Washout (7 Days), CLP (7 Days): Subjects in this group received coadministration of CLP orally and spironolactone orally in Period 1/administration of CLP orally alone in Period 2.
- CLP (7 Days), Washout (7 Days), CLP + Spiro (7 Days): Subjects in this group received administration of CLP alone orally in Period 1/coadministration of CLP orally and spironolactone orally in Period 2.
Period: Period 1
Arm/Group | CLP + Spiro (7 Days), Washout (7 Days), CLP (7 Days) | CLP (7 Days), Washout (7 Days), CLP + Spiro (7 Days)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | CLP + Spiro (7 Days), Washout (7 Days), CLP (7 Days) | CLP (7 Days), Washout (7 Days), CLP + Spiro (7 Days)
Started | 8 (1 subject discontinued during the washout period prior to starting treatment period 2.) | 9
Completed | 7 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CLP + Spiro/CLP: Subjects in this group received coadministration of CLP orally and spironolactone orally in Period 1/administration of CLP orally alone in Period 2.
- CLP/CLP + Spiro: Subjects in this group received administration of CLP alone orally in Period 1/coadministration of CLP orally and spironolactone orally in Period 2.
- Total: Total of all reporting groups
Arm/Group | CLP + Spiro/CLP | CLP/CLP + Spiro | Total
Number analyzed (Participants) | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (7.58) | 63.4 (9.77) | 59.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 8 | 13
Weight [Mean (Standard Deviation); unit: kg] | 91.35 (24.20) | 99.54 (27.49) | 95.4 (25.8)
Diet [Number; unit: participants]
  Low sodium | 1 | 2 | 3
  Medium sodium | 1 | 1 | 2
  High sodium | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Fecal Sodium Content
Description: Change =(Days 10-13/29-32 Daily Average)-(Days 3-6/22-25 Daily Average)
Time Frame: baseline average (days 3-6 or days 22-25) and treatment average (days 10-13 or 29-32)
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Treatment Group: CLP Alone: oral administration
- Treatment Group: CLP + Spironolactone: CLP: oral administration Spironolactone: oral administration
Arm/Group | Treatment Group: CLP Alone | Treatment Group: CLP + Spironolactone
Number analyzed (Participants) | 16 | 18
mg | 635.10 (441.11) | 501.95 (342.52)
Statistical Analysis 1: Comparison: Treatment Group: CLP Alone vs Treatment Group: CLP + Spironolactone; One-way analysis of covariance (ANCOVA) common slopes model for a 2-period crossover design; Test type: Superiority or Other; p = 0.0662, ANCOVA

2. Secondary Outcome: Change in Fecal Weight
Description: Change = (Days 10-13/29-32 Daily Average) - (Days 3-6/22-25 Daily Average)
Time Frame: baseline average (days 3-6 or 22-25) and treatment average (days 10-13 or 29-32)
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Treatment Group: CLP Alone: CLP: oral administration
Arm/Group | Treatment Group: CLP Alone | Treatment Group: CLP + Spironolactone
Number analyzed (Participants) | 16 | 18
grams | 144.7 (86.50) | 119.0 (106.98)
Statistical Analysis 1: Comparison: Treatment Group: CLP Alone vs Treatment Group: CLP + Spironolactone; One-way analysis of covariance (ANCOVA) common slopes model for a 2-period crossover design; Test type: Superiority or Other; p = 0.1899, ANCOVA

ADVERSE EVENTS:
Arm/Group | Treatment Group: CLP Alone | Treatment Group: CLP + Spironolactone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 5/16 | 8/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: CLP Alone (N=16) | Treatment Group: CLP + Spironolactone (N=18)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotenstion (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other